CLINICAL TRIAL: NCT05235984
Title: Technical Feasibility Study on Screening Sleep Related Breathing Disturbances and Sleep Apnoea With Wearable Sensors
Acronym: Screenbeat
Status: Completed | Type: Observational
Sponsor: Firstbeat Technologies Oy (Industry)
Collaborators: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Responsible Party: Sponsor
Other Study IDs: Screenbeat_SA
Record Dates: First submitted 2022-02-10; First posted 2022-02-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Sleep Apnea; Sleep Disorder
Keywords: apnea; apnoea; sleep
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Wake Disorders; Apnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the feasibility of detecting sleep apnoeas with unobtrusive wearable sensors and sounds recorded with a smartphone is studied by making an overnight recording to patients with high probability of sleep apnoeas. The data acquired with the aforementioned devices is: ECG, acceleration, bioimpedance of thorax and processed and raw audio. In data analysis phase it will be studied which combinations of these signals would enable detecting sleep apnoeas with high enough sensitivity and specificity when compared to a night polygraphy reference (Nox T3 device using airflow, breathing movements, audio, position, movement, oxygen saturation, pulse and leg EMG).

ELIGIBILITY:
Inclusion Criteria:

* High a priori probability for SA based on previous PG findings, BMI, and ESS and medical history
* Clinical reason i.e. potential benefit of repeating the PG due to e.g. technical challenges in the previous PG and/or unclear findings or diagnosis. Participation may be offered also in cases where first PG is diagnostic. In these cases accuracy of sleep apnoea grading will be improved.
* Adequate Finnish language skills to comprehend study-related instructions and questionnaires. The study materials are available only in Finnish.
* Signed written informed consent

Exclusion Criteria:

* Medical history of a major cardiovascular event (myocardial infarction, coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), stroke, or transient ischemic attack) within the previous 6 months
* Use of cardiac pacemaker or history of atrial fibrillation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group will be recruited from occupational health care patients who have been earlier admitted by Mehiläinen for a PG study at KNF-laboratoriot.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of apnoea detection using the Screenbeat technology | 1 day
  The sensitivity and specificity of apnoea detection using the Screenbeat technology with different combinations of electrocardiogram (ECG), movement, bioimpedance and audio data, as measured by the AHI (apnoea-hypopnoea events per hour). The clinical reference for SA detection will be provided by PG.

CONTACTS AND LOCATIONS:
Overall Officials: Juha K Heiskala, LM, DSc, Study Director — Neurophysiologist at HUS (Hospital district of Helsinki and Uusimaa) and at KNF-Laboratoriot Oy; Ilkka Korhonen, DSc, Principal Investigator — CTO at Firstbeat Technologies and Associate Professor at Tampere University
Locations (1):
- KNF-Laboratoriot Oy, Helsinki, Southern Finland, Finland